CLINICAL TRIAL: NCT05502926
Title: Perioperative Lung Ultrasound Score (LUS) for Prediction of Postoperative Pulmonary Complications (PPC)
Brief Title: Use of Point-of-care Lung Ultrasound Before and After Surgery Trying to Predict Post-operative Pulmonary Complications
Status: Completed | Type: Observational
Sponsor: Moshe Rucham MD (Other)
Responsible Party: Sponsor-Investigator, Moshe Rucham MD, Principal Investigator, Soroka University Medical Center
Organization: Soroka University Medical Center (Other)
Other Study IDs: SOR001022CTIL
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ultrasonography; Postoperative Complications; Anesthesia; Surgery-Complications; Pulmonary Complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lung ultrasound score — peroperative and postoperative 12 point trans-thoracic lung ultrasound

SUMMARY:
Patients undergoing surgery inside their abdomen, with no serious heart or lung diseases, will have a lung ultrasound exam before and after surgery. The patient respiratory status in the post-operative unit and the surgical ward will be monitored for complications after surgery

DETAILED DESCRIPTION:
The study will be performed in the Soroka hospital operating room and recovery unit.

On admission to pre-surgery, patients will be investigates for inclusion and exclusion criteria. Those that are eligible for the study will be asked to give formal consent to participate in the study. After consent the examiner will review the patient's past medical history and surgery plan, and will preform the pre-operative LUS exam.

After surgery, the examiner will review the electronic anesthesia record and will preform the post-operative LUS exam within 30 minutes of arrival to the recovery unit or 30 minutes from extubation (in patients that were admitted to the recovery unit still under mechanical ventilation). Upon discharge from the recovery unit the examiner will review the recovery unit electronic record.

After discharge, the examiner will review the patient post-operative surgical ward electronic record.

ELIGIBILITY:
Inclusion Criteria:

The population study will include patients 18 years and older, with ASA class I, II or III, presenting for elective intra-abdominal surgery under general anesthesia and are not planned for long-term post-surgical mechanical ventilation.

Exclusion Criteria:

Patient will be excluded from the study if they have pre-existing moderate or severe heart or lung disease: a history of ischemic heart disease, moderate or severe systolic or diastolic heart failure, moderate or severe pulmonary hypertension, moderate or severe obstructive or interstitial lung disease. Patients will also be excluded if they had a severe intra-operative pulmonary complication (laryngospasm, bronchospasm, anaphylaxis, emergency surgical airway). Patients who require un-planned long term mechanical ventilation or those who died during surgery will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients presented for elective intra-abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
post operative oxygen treatment | 48 hours
  any kind of oxygen therapy (face mask, nasal cannula, CPAP/BIPAP) more then 12 hours after and of surgery, or desaturation <90%
icu admission / reintubation | during hospital stay
  unplanned postoperative admission to icu or re-intubation
postoperative pneumonia | 48 hours
  clinical or radiographic diagnosis of pneumonia
death | 48 hours
  postoperative death of any cause

SECONDARY OUTCOMES:
PACU stay | during hospital stay
  total length of stay at the post operative care unit
PACU oxygen therapy | during hospital stay
  total time with oxygen treatment (nasal cannula, face mask) in the post operative care unit
PACU discharge oxygen therapy | during hospital stay
  oxygen treatment (nasal cannula, face mask) on discharge from the post operative care unit

CONTACTS AND LOCATIONS:
Overall Officials: evgeni brotfaine, prof, Study Director — Soroka University Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Undecided
this is a preliminary study in this subject

REFERENCES:
- [Derived] Rucham M, Lior Y, Fuchs L, Gruenbaum BF, Acker A, Zlotnik A, Brotfain E. Perioperative Lung Ultrasound Findings in Elective Intra-Abdominal Surgery: Associations with Postoperative Pulmonary Complications. J Clin Med. 2024 Nov 24;13(23):7098. doi: 10.3390/jcm13237098. PMID 39685557